CLINICAL TRIAL: NCT04649658
Title: Awake Prone Position in Critical and Severe COVID-19 Patients Undergoing Noninvasive Respiratory Support: a Retrospective Multicenter Cohort Study
Brief Title: Pronation in COVID-19 Patients Undergoing Non Invasive Respiratory Support
Acronym: PRINCESS
Status: Completed | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Roberto Tonelli, MD, University of Modena and Reggio Emilia
Other Study IDs: UModenaReggio10
Record Dates: First submitted 2020-11-30; First posted 2020-12-02 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Covid19
Keywords: Spontaneous breathing; Awake pronation; COVID-19; Respiratory failure
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency | interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prone position: Severe and critical COVID-19 patients undergoing non invasive respiratory support subjected to prone position
  Interventions: Behavioral: Prone position
- Standard care: Severe and critical COVID-19 patients undergoing non invasive respiratory support subjected to standard care

INTERVENTIONS:
Behavioral: Prone position — Prone position maintained at least 3 hours/day
  Groups: Prone position

SUMMARY:
Pronation seems feasible and effective in improving blood oxygenation in patients with COVID-19 pneumonia. Data are lacking on the effects of pronation on clinical outcome in this subset of patients.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

* patients aged ≥18 and < 80 years old
* acute respiratory failure

Exclusion Criteria:

* endotracheal intubation performed within the first 24 hours from admission,
* ceiling of escalation of intensive care
* do not intubate order as expressed by patient willing or upon clinical judgement
* missing core data at medical record analysis (clinical features at baseline, pronation information, type and time of ventilatory support required, mortality, need for tracheostomy, length of respiratory intensive care unit and hospital stay).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients aged ≥18 and < 80 years old admitted to the two respiratory intensive care units for severe and critical COVID-19 pneumonia between March 1st, 2020 and June 1st, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Endotracheal intubation | 28 days

SECONDARY OUTCOMES:
Mortality | 28 days
Tracheostomy | 28 days
Length of Respiratory Intensive Care Unit stay | 60 days
Length of Hospital stay | 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Policlinico di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: No